CLINICAL TRIAL: NCT04797169
Title: Noom Health for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Noom Inc. (Industry)
Responsible Party: Principal Investigator, Tom Hildebrandt, Associate Professor and Chief of the Division of Eating & Weight Disorders, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-2224
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Weight Loss; Obesity
Keywords: Weight Loss; Mobile App; Digital Health; Weight Loss Maintenance; Weight Loss Suppression; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions in a parallel design including a 12-month intervention. Participants will be openly-enrolled over the course of 12-months until the recruitment goal of 600, 300 in each group, is reached.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noom Health (Experimental)
  Interventions: Behavioral: Noom Health
- Noom Digital Health (Active Comparator)
  Interventions: Behavioral: Noom Digital Health

INTERVENTIONS:
Behavioral: Noom Health — In Noom Health, participants will be encouraged to use the Noom app multiple times a day to log eating episodes, physical activity and weight. They will also have the ability to interact with coaches to receive advice and feedback specific to weight loss.
  Arms: Noom Health
Behavioral: Noom Digital Health — In Noom Digital Health, participants will use a simplified version to log eating episodes and weight. Both conditions will receive the same weight loss advice content.
  Arms: Noom Digital Health

SUMMARY:
The goals of the study are to use the Noom mobile app to help individuals with weight loss and weight loss maintenance. This project will test the comparative efficacy of Noom Health vs. Noom Digital Health for weight loss, quality of life, psychosocial functioning, and self-reported health status. It is expected that use of Noom Health will show post-intervention success relative to Noom Digital Health as well as long-term success with weight loss maintenance. Data is expected to show that participants who are older, have less support, have more health conditions, and with more psychosocial problems will benefit more from Noom Health. It is also expected that confidence in the ability to lose weight will produce more successful results in Noom Health vs. Noom Digital Health.

DETAILED DESCRIPTION:
A total of 600 subjects will be enrolled in a randomized-controlled trial comparing the Noom app (Noom Health) to a digital control (Noom Digital Health) with 6 months of intervention and 6 months active maintenance in both groups. Measures will include demographics, psychosocial measures, height/weight, waist circumference, weight loss history/practices, health care practices/utilization, and quality of life.

Participants will complete informed consent and interviews via a HIPAA-compliant videoconference (Zoom) and other questionnaires via a REDCap interface. All participants will complete screening/baseline procedures to determine eligibility and initial information. Subsequently, they will be randomized to one of the groups for a 6-month intervention and 6- month maintenance period (12 months total).

In Noom Health, participants will be encouraged to use the app multiple times per day to log eating episodes, physical activity and weight. Coaches will also interact with participants directly through the app. In Noom Digital Health, participants will use a simplified version to log eating episodes and weight. Both conditions will receive the same weight loss advice content.

During the intervention, participants will complete monthly satisfaction surveys. Additionally, follow-up measures will be conducted at 7 time points (Screening/Baseline, 1 month, 4 months, 6 months, 12 months, 18 months, 24 months, and 30 months).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be interested in the Noom app
* BMI > 27 kg/m2
* Ages of 18 and 60 at entry to the study
* Speak English

Exclusion Criteria:

* Contraindication to smartphone use (e.g., seizures from prior smartphone use, do not own a smartphone)
* Acute suicide risk
* Pregnant or planning to become pregnant during the study
* Current Noom use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Psychiatry, Eating and Weight Disorders Program, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sysko R, Bibeau J, Boyar A, Costello K, Michaelides A, Mitchell ES, Susanin A, Hildebrandt T. A 2.5-Year Weight Management Program Using Noom Health: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 12;11(8):e37541. doi: 10.2196/37541. PMID 35969439

RESULTS

PARTICIPANT FLOW:
Groups:
- Noom Health: In Noom Health, participants encouraged to use the Noom app multiple times a day to log eating episodes, physical activity and weight. They will also have the ability to interact with coaches to receive advice and feedback specific to weight loss.
- Noom Digital Health: In Noom Digital Health, participants used a simplified version to log eating episodes and weight. Both conditions will receive the same weight loss advice content.
Period: Overall Study
Arm/Group | Noom Health | Noom Digital Health
Started | 302 | 298
Completed | 190 | 193
Not Completed | 112 | 105
Not completed — Lost to Follow-up | 84 | 67
Not completed — Pregnancy | 1 | 3
Not completed — Withdrawal by Subject | 27 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Noom Health | Noom Digital Health | Total
Number analyzed (Participants) | 302 | 298 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9) | 42 (9) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 246 | 497
  Male | 51 | 52 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 277 | 274 | 551
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 260 | 249 | 509
  More than one race | 14 | 15 | 29
  Unknown or Not Reported | 5 | 6 | 11
Weight [Mean (Standard Deviation); unit: pounds] | 210.1 (42.1) | 211.7 (44.7) | 210.9 (43.4)
24-hr Caloric Intake [Mean (Standard Deviation); unit: calories] — Caloric Intake using the Automated Self-Administered Recall System (ASA24)
  calories | 2186.6 (957.3) | 2118.2 (908.1) | 2152.7 (933.0)
EDEQ Global [Mean (Standard Deviation); unit: units on a scale] — Dietary Behavior assessed by the Eating Disorder Examination Questionnaire (EDE-Q) global score. Dietary restraint, eating, shape, and weight concerns are measured with the EDE-Q. These subscales are summed and then divided by the total number of subscales (4) to create a global score. Scores range from 0 to 52 with higher scores indicating higher severity.
  units on a scale | 2.5 (0.9) | 2.6 (1.0) | 2.5 (1.0)
Metabolic Equivalents (METS) Value measured by IPAQ [Mean (Standard Deviation); unit: METS Value] — Physical Activity using the International Physical Activity Questionnaire (IPAQ). The IPAQ includes 27 items and determines a MET value for time spent in an average week completing different levels of activity including vigorous or moderate physical activity, walking, and sitting. One MET is the energy spent sitting at rest.
  METS Value | 2328.1 (1638.2) | 2249.0 (1577.6) | 2288.8 (1607.5)
The Depression Anxiety Stress Scales (DASS) [Mean (Standard Deviation); unit: units on a scale] — DASS a 42-item self-report scale of negative emotional states with subscales of depression, anxiety, and stress. Each subscale is scored 0-42, with total score from 0-126. Higher scores indicate more severe psychological distress.
  units on a scale
    Depression | 4.5 (5.4) | 5.0 (5.9) | 4.7 (5.6)
    Anxiety | 2.8 (3.9) | 3.1 (3.8) | 3.0 (3.8)
    Stress | 7.8 (6.8) | 8.6 (7.4) | 8.2 (7.1)
Sleep Impairment using the PROMIS Sleep Related Impairment Survey Sleep impairment [Mean (Standard Deviation); unit: t-score] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment v.1.0 is a 16-item self-report measure of perceived functioning during waking hours in relation to tiredness and trouble sleeping. A raw score is calculated by summing all individual items and is translated into a T-score with standard error (SE). A T-score of 50 indicates normal impairment compared to the general population, scores above 50 indicate more impairment.
  t-score | 35.7 (11.7) | 37.5 (11.8) | 36.6 (11.8)
Short Form 36 (SF-36) [Mean (Standard Deviation); unit: units on a scale] — The Short-Form-36 (SF-36) is a 36-item self-report health-related quality of life assessment of physical functioning, limitations, energy, emotional well-being, social functioning, pain and general health.
  Physical Composite Score (PCS) range from 17.2- 66.7 with lower scores indicating worse quality of life related to physical health.
  Mental Composite Score (MCS) range from 12.7-64.2 with lower scores indicating worse quality of life related to mental health.
  units on a scale
    Physical Composite | 43.1 (10.2) | 42.3 (1.03) | 42.7 (10.3)
    Mental Composite | 53.4 (7.2) | 53.1 (7.5) | 53.3 (7.4)
Self-Efficacy for Healthy Eating using the Diet Self-Efficacy Scale (DIET-SE) [Mean (Standard Deviation); unit: units on a scale] — Self-Efficacy for Healthy Eating using the Diet Self-Efficacy Scale (DIET-SE) is an 11-item self-report assessment of healthy eating with scales specific to temptations, social/internal factors, and negative emotional related to resistance. The score ranges from 0 - 40 with higher scores indicating more self-efficacy.
  units on a scale | 16.3 (9.6) | 16.4 (9.5) | 16.4 (9.6)
CDC NCHS National Health Interview Survey [Mean (Standard Deviation); unit: visits/months] — Using an adapted version of the CDC National Center for Health Statistics (NCHS) National Health Interview Survey, the survey includes 4 questions about healthcare utilization. Items identify type of healthcare sought and frequency. The frequency of provider visits will be calculated to determine healthcare utilization. A frequency score of zero indicates no healthcare utilized. There is no upper limit for the frequency.
  visits/months | 1.8 (2.4) | 1.7 (3.6) | 1.7 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline
Description: Weight at 6 months and 30 months as compared to baseline. Weight will be documented using staff-led Zoom calls and taken with the participant's home scale.
Time Frame: Baseline, 6 months and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
lbs
  Baseline | 210.1 (42.1) | 211.7 (44.7)
  6 months: number analyzed (Participants) | 236 | 231
  6 months | 199.4 (41.4) | 204.6 (45.8)
  30 months: number analyzed (Participants) | 190 | 193
  30 months | 197.2 (43.1) | 201.6 (43.6)

2. Secondary Outcome: Change in Caloric Intake Using the Automated Self-Administered Recall System (ASA24) From Baseline to 30 Months
Description: Caloric intake at 30 months as compared to baseline. Caloric intake will be measured using the ASA24 dietary recall system.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
calories
  Baseline | 2186.6 (957.3) | 2118.2 (908.1)
  30 months: number analyzed (Participants) | 106 | 112
  30 months | 1681.7 (906.9) | 1578.5 (784.8)

3. Secondary Outcome: Change in Dietary Behavior Using the Eating Disorder Examination Questionnaire (EDE-Q) From Baseline to 30 Months
Description: EDE-Q global score at 30 months as compared to baseline. Dietary restraint, eating, shape, and weight concerns are measured with the EDE-Q. These subscales are summed and then divided by the total number of subscales (4) to create a global score. Scores range from 0 to 52 with higher scores indicating higher severity.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 2.5 (0.9) | 2.6 (1.0)
  30 months: number analyzed (Participants) | 119 | 123
  30 months | 1.7 (1.1) | 1.8 (1.2)

4. Secondary Outcome: Change in Physical Activity Using the International Physical Activity Questionnaire (IPAQ) From Baseline to 30 Months
Description: Physical activity at 30 months as compared to baseline. The IPAQ includes 27 items and determines a MET value for time spent in an average week completing different levels of activity including vigorous or moderate physical activity, walking, and sitting. One MET is the energy spent sitting at rest.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: Met Value
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
Met Value
  Baseline | 2328.1 (1638.2) | 2249.0 (1577.6)
  30 months: number analyzed (Participants) | 118 | 122
  30 months | 1919.6 (1463.0) | 1973.9 (1748.8)

5. Secondary Outcome: Change in Depression Using the Depression Anxiety Stress Scales (DASS) From Baseline to 30 Months
Description: Depression subscale score at 30 months as compared to baseline. DASS is a 42-item self-report scale of negative emotional states with subscales of depression, anxiety, and stress. Each subscale is scored 0-42, with total score from 0-126. Higher scores indicate more severe psychological distress.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 4.5 (5.4) | 5.0 (5.9)
  30 months: number analyzed (Participants) | 117 | 121
  30 months | 3.9 (7.2) | 4.4 (6.8)

6. Secondary Outcome: Change in Anxiety Using the Depression Anxiety Stress Scales (DASS) From Baseline to 30 Months
Description: Anxiety subscale score at 30 months as compared to baseline. DASS is a 42-item self-report scale of negative emotional states with subscales of depression, anxiety, and stress. Each subscale is scored 0-42, with total score from 0-126. Higher scores indicate more severe psychological distress.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 2.8 (3.9) | 3.1 (3.8)
  30 months: number analyzed (Participants) | 117 | 121
  30 months | 2.4 (4.8) | 2.7 (4.4)

7. Secondary Outcome: Change in Stress Using the Depression Anxiety Stress Scales (DASS) From Baseline to 30 Months
Description: Stress subscale score at 30 months as compared to baseline. DASS a 42-item self-report scale of negative emotional states with subscales of depression, anxiety, and stress. Each subscale is scored 0-42, with total score from 0-126. Higher scores indicate more severe psychological distress.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 7.8 (6.8) | 8.6 (7.4)
  30 months: number analyzed (Participants) | 117 | 121
  30 months | 5.4 (7.3) | 6.7 (8.3)

8. Secondary Outcome: Change in Sleep Impairment Using the PROMIS Sleep Related Impairment Survey From Baseline to 30 Months
Description: Sleep impairment at 30 months as compared to baseline. The PROMIS Sleep Related Impairment v.1.0 is a 16-item self-report measure of perceived functioning during waking hours in relation to tiredness and trouble sleeping. A raw score is calculated by summing all individual items and is translated into a T-score with standard error (SE). A T-score of 50 indicates normal impairment compared to the general population, scores above 50 indicate more impairment.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
t-score
  Baseline | 35.7 (11.7) | 37.5 (11.8)
  30 months: number analyzed (Participants) | 117 | 120
  30 months | 31.6 (11.6) | 33.9 (12.4)

9. Secondary Outcome: Change in Physical Composite Score (PCS) Using the Short-Form-36 (SF-36) From Baseline to 30 Months
Description: PCS at 30 months as compared to baseline. The SF-36 is a 36-item self-report health-related quality of life assessment of physical functioning, limitations, energy, emotional well-being, social functioning, pain and general health. Scores range from 17.2- 66.7 with lower scores indicating worse quality of life related to physical health.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 43.1 (10.2) | 42.3 (10.3)
  30 months: number analyzed (Participants) | 116 | 120
  30 months | 45.9 (10.1) | 44.8 (11.4)

10. Secondary Outcome: Change in Mental Composite Score (MCS) Using the Short-Form-36 (SF-36) From Baseline to 30 Months
Description: MCS at 30 months as compared to baseline. The SF-36 is a 36-item self-report health-related quality of life assessment of physical functioning, limitations, energy, emotional well-being, social functioning, pain and general health. Scores range from 12.7-64.2 with lower scores indicating worse quality of life related to mental health.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 53.4 (7.2) | 53.1 (7.5)
  30 months: number analyzed (Participants) | 116 | 120
  30 months | 53.5 (7.6) | 54.9 (7.4)

11. Secondary Outcome: Change in Self-Efficacy for Healthy Eating Using the Diet Self-Efficacy Scale (DIET-SE) From Baseline to 30 Months
Description: Self-efficacy at 30 months as compared to baseline. The DIET-SE is an 11-item self-report assessment of healthy eating with scales specific to temptations, social/internal factors, and negative emotional related to resistance. The score ranges from 0 - 40 with higher scores indicating more self-efficacy.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
score on a scale
  Baseline | 16.3 (9.6) | 16.4 (9.5)
  30 months: number analyzed (Participants) | 115 | 120
  30 months | 23.0 (11.4) | 21.7 (12.9)

12. Secondary Outcome: Adherence to Intervention Measured Using a Percentage of the Total Number of Available App Features Used at 6 Months
Description: The percent of available features on the app, expected verses completed at 6 months
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of available features on app
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
percentage of available features on app | 38.4 (24.2) | 17.9 (15.2)

13. Secondary Outcome: Number of Participants With 12-Month Completion Status
Description: Attrition at 12 months as compared to number randomized at baseline documented using completion status
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
Participants | 220 | 222

14. Secondary Outcome: Percent of Successful Technological Fixes
Description: App compatibility will be examined by calculating the percent of successful technological fixes at 12 months as compared to baseline. The type of technological problems encountered by participants while using the app and any fixes needed will be categorized.
Time Frame: Baseline and 12 Months
Measure: Number; unit: percent of successful tech fixes
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
percent of successful tech fixes | 86 | 81

15. Secondary Outcome: Change in CDC NCHS National Health Interview Survey
Description: Changes in health status from baseline to 30-months as measured by questions from the CDC NCHS National Health Interview Survey. Using an adapted version of the CDC NCHS National Health Interview Survey, the survey includes 4 questions about healthcare utilization. Items identify type of healthcare sought and frequency. The frequency of provider visits will be calculated to determine healthcare utilization. A frequency score of zero indicates no healthcare utilized. There is no upper limit for the frequency.
Time Frame: Baseline and 30 Months
Population: Results available for participants who had study visit and provided data.
Measure: Mean (Standard Deviation); unit: visits/months
Arm/Group | Noom Health | Noom Digital Health
Number analyzed (Participants) | 302 | 298
visits/months
  Baseline | 1.8 (2.4) | 1.7 (3.6)
  30 months: number analyzed (Participants) | 119 | 122
  30 months | 1.9 (3.0) | 1.8 (3.0)

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Noom Health | Noom Digital Health
All-Cause Mortality (participants affected / at risk) | 0/302 | 0/298
Serious Adverse Events (participants affected / at risk) | 1/302 | 2/298
Other Adverse Events (participants affected / at risk) | 43/302 | 42/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noom Health (N=302) | Noom Digital Health (N=298)
Breastfeeding supply lowered (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Fainted during exercise (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noom Health (N=302) | Noom Digital Health (N=298)
Colitis - unrelated (Gastrointestinal disorders) | 0 | 1
Food poisoning - unrelated (Gastrointestinal disorders) | 1 | 0
Stomach cramps - unrelated (Gastrointestinal disorders) | 0 | 1
Allergic reaction - unrelated (General disorders) | 1 | 0
Dental problem - unrelated (General disorders) | 0 | 1
Unknown health problem - unrelated (General disorders) | 2 | 0
Viral/bacterial Illness - unrelated (Infections and infestations) | 19 | 16
Car accident - unrelated (Injury, poisoning and procedural complications) | 0 | 1
Injury - unrelated (Injury, poisoning and procedural complications) | 2 | 2
Fibromyalgia - unrelated (Musculoskeletal and connective tissue disorders) | 1 | 0
Multiple Sclerosis - unrelated (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain/muscular issue - unrelated (Musculoskeletal and connective tissue disorders) | 3 | 1
Cancer - unrelated (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breastfeeding - unrelated (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy - unrelated (Pregnancy, puerperium and perinatal conditions) | 7 | 10
Anxiety - unrelated (Psychiatric disorders) | 1 | 1
Depression - unrelated (Psychiatric disorders) | 0 | 1
Swelling - unrelated (Skin and subcutaneous tissue disorders) | 1 | 1
Surgery - unrelated (Surgical and medical procedures) | 2 | 3
Migraine - unrelated (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT04797169/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04797169/ICF_001.pdf